CLINICAL TRIAL: NCT00574002
Title: Defining the Threshold for Safe Chest Tube Removal.
Brief Title: Establishing Safe Drainage Limits for Pleural Chest Tube Removal.
Status: Withdrawn | Type: Observational
Why Stopped: Low study enrollment; re-evaluating study protocol and study selection criteria.
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 07-68e
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Thoracic Surgery; Thoracic Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients that have their chest tube removed when drainage is 400mL or less in 24 hours.
- Group B.: Patients that have their chest tube removed when drainage is 200mL or less in 24 hours.

SUMMARY:
The purpose of the study is to evaluate a safe threshold for when to remove chest tubes in patients based on the amount of drainage present.

DETAILED DESCRIPTION:
Measurement of pleural fluid drainage in chest tubes of trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one chest tube
* No air leak present
* Fluid is not infected
* Pleural drainage of fluid was an indication for placement of the chest tube
* Patient is post-thoracic surgery
* Patient is post-thoracic trauma
* Informed consent obtained

Exclusion Criteria:

* Presence of air leak
* Infected pleural fluid
* Active intra-thoracic bleeding
* Thoracic empyema
* Non-removal of chest tube (i.e.: expired)
* Pregnancy
* Less than 18 years of age
* Unable to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Repeat chest tube insertion within 30 days | two years
Thoracotomy on affected side within 30 days | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Gerald L. Early, M.D., M.A., Principal Investigator — Truman Medical Center
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States